CLINICAL TRIAL: NCT05882058
Title: DAREON™-5: An Open-label, Multi-center Phase II Dose Selection Trial of Intravenous BI 764532, a DLL3-targeting T Cell Engager, in Patients With Relapsed/Refractory Extensive-stage Small Cell Lung Cancer and in Patients With Other Relapsed/Refractory Neuroendocrine Carcinomas
Brief Title: DAREON™-5: A Study to Test Whether Different Doses of BI 764532 Help People With Small Cell Lung Cancer or Other Neuroendocrine Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1438-0005; 2023-504247-13-00 (Registry Identifier: CTIS); U1111-1292-4406 (Registry Identifier: UTN, WHO registry)
Record Dates: First submitted 2023-05-22; First posted 2023-05-31 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Small Cell Lung Carcinoma; Neuroendocrine Neoplasms; Extra-pulmonary Neuroendocrine Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: The trial consists of 2 parts:
  Part 1: open label, randomized, with 2 treatment arms followed by Part 2: open label, non-randomized, 1 treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose group 1 (Experimental)
  Interventions: Drug: BI 764532, dose 1
- Part 1: Dose group 2 (Experimental)
  Interventions: Drug: BI 764532, dose 2
- Part 2: Expansion cohort (Experimental)
  Interventions: Drug: BI 764532, dose 1

INTERVENTIONS:
Drug: BI 764532, dose 1 — BI 764532, dose 1
  Other Names: Obrixtamig
  Arms: Part 1: Dose group 1; Part 2: Expansion cohort
Drug: BI 764532, dose 2 — BI 764532, dose 2
  Other Names: Obrixtamig
  Arms: Part 1: Dose group 2

SUMMARY:
This study is open to adults with small cell lung cancer and other neuroendocrine tumours. The study is in people with advanced cancer for whom previous treatment was not successful or no standard treatment exists.

The purpose of this study is to find a suitable dose of BI 764532 that people with advanced cancer can tolerate. 2 different doses of BI 764532 are tested in this study. Another purpose is to check whether BI 764532 can make tumours shrink. BI 764532 is an antibody-like molecule (DLL3/CD3 bispecific) that may help the immune system fight cancer.

The study has 2 parts. In Part 1, participants are put into 2 groups randomly, which means by chance. Participants have an equal chance of being in either group. One group gets dose 1 of BI 764532 and the other group gets dose 2 of BI 764532. In Part 2, all participants receive the same dose of BI 764532. Part 2 is open to people with a certain kind of tumour called extrapulmonary neuroendocrine carcinoma.

All participants receive BI 764532 as an infusion into a vein when starting treatment. If there is benefit for the participants and if they can tolerate it, the treatment is given up to the maximum duration of the study. During this time, participants visit the study site regularly. The total number of visits depends on how they respond to and tolerate the treatment.

The first study visits include an overnight stay to monitor participants´ safety. Doctors record any unwanted effects and regularly check the general health of the participants.

ELIGIBILITY:
Inclusion criteria:

1. Male or female participants ≥18 years old and at least at the legal age of consent in countries where it is greater than 18 years at the time of signature of the informed consent form (ICF).
2. Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
3. Part 1: Histologically or cytologically confirmed, cancer of the following histologies:

   * Small cell lung cancer (SCLC)
   * Extra-pulmonary neuroendocrine carcinoma (epNEC) (except Merkel cell carcinoma (MCC), Medullary thyroid cancer (MTC) and Neuroendocrine prostate cancer (NEPC))
   * Large cell neuroendocrine carcinoma (LCNEC) of the lung Patients with tumours with mixed histologies for any above type are eligible only if the neuroendocrine carcinoma/small tumour cells component is predominant and represents at least 50% of the overall tumour tissue.

   Patients must have progressed or recurred after standard of care therapy
   * SCLC: after at least two prior lines of therapy, including at least one platinum-based regimen; in countries where standard of care in first line therapy includes PD-L1 inhibitor treatment patients should have received the combination of platinum-based regimen plus PD-L1 inhibitor unless they have been unable to receive checkpoint inhibitor treatment.
   * Therapy includes PD-L1 inhibitor treatment; patients should have received the combination of platinum-based regimen plus PD-L1 inhibitor unless they have been unable to receive checkpoint inhibitor treatment.

     * epNEC/LCNEC: after at least one platinum-based regimen. Part 2: Histologically or cytologically confirmed epNEC (except MCC, MTC and NEPC) with centrally assessed DLL3 high expression status. Patients must have progressed or recurred after at least one platinum-based regimen.
4. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
5. Measurable lesions as defined per Response Evaluation Criteria In Solid Tumours (RECIST) v 1.1 within 21 days prior to the first dose of BI 764532.
6. Part 1: Availability of archival tumour tissue sample Part 2: Availability of archival formalin-fixed paraffin-embedded (FFPE) tumour tissue sample. Following specimens are not allowed: Fine Needle Aspiration (FNA), Cytology samples, decalcified bone samples.
7. Adequate organ function as defined in the protocol.
8. All toxicities related to previous anti-cancer therapies have resolved = Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 prior to trial treatment administration (except for alopecia, peripheral neuropathy, fatigue and endocrinopathies controlled by replacement therapy which must be = CTCAE Grade 2 and amenorrhea/menstrual disorders which can be any grade).
9. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of their use is provided in the participant information

Exclusion criteria:

1. Untreated or symptomatic brain metastases. (Part 2: with mandatory assessment by brain MRI within 21 days before first trial drug administration.) Participants with treated, stable brain metastases are eligible provided they meet the following criteria:

   * Radiotherapy or surgery for brain metastases was completed at least 2 weeks prior to the first administration of BI 764532.
   * Patient is off steroids for at least 7 days (physiologic doses of steroids are permitted), and the patient is off anti-epileptic drugs for at least 7 days or on stable doses of anti-epileptic drugs for malignant central nervous system (CNS) disease.
2. Presence of leptomeningeal disease or, part 2: epidural disease including spinal cord compression.
3. Part 1: Active/previous history of interstitial lung disease or non-infectious pneumonitis (any grade).

   Part 2: Active/previous history of interstitial lung disease, pulmonary fibrosis, organizing pneumonia or non-infectious pneumonitis (any grade). Patients with a history of therapy-related pneumonitis that is considered clinically resolved are eligible.
4. Participants who experienced severe, life-threatening immune-mediated adverse events or infusion-related reactions including those that lead to permanent discontinuation while on treatment with immuno-oncology agents.
5. Prior anti-cancer therapy:

   * Patients who have been treated with any other anti-cancer drug within 4 weeks or within 5 half-life periods (whichever is shorter) prior to first administration of BI 764532.
   * Patients who have been treated with extensive field radiotherapy including whole brain irradiation within 2 weeks prior to first administration of BI 764532.
6. Previous treatment with Delta-like ligand 3 (DLL3)-targeting T cell engagers or cell therapies.
7. Diagnosis of immunodeficiency or systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of BI 764532. Physiological replacement of steroids is allowed.
8. Unresolved toxicity from prior anti-tumour therapy, defined as per protocol. Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-02-24 (Estimated)

PRIMARY OUTCOMES:
Part 1: Objective response (OR), defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) | up to 26 months
  according to RECIST v 1.1 by investigator assessment from the date of treatment start until the earliest date of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Part 1: Occurrence of treatment-emergent adverse events (TEAEs) during the on-treatment period | up to 26 months
Part 2: Objective response (OR) | up to 27 months
  Objective response is defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST v 1.1 by blinded independent central review from the date of treatment start until the earliest date of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent

SECONDARY OUTCOMES:
Part 1: Duration of objective response (DOR) based on investigator assessment | up to 26 months
  DOR is defined as the time from first documented confirmed OR until the earliest date of disease progression or death among patients with confirmed OR.
Part 1: Progression-free survival (PFS) based on investigator assessment | up to 26 months
  PFS is defined as the time from treatment start until the earliest date of tumour progression according RECIST v 1.1 or death from any cause, whichever occurs first.
Part 1: Disease control (DC), defined as best overall response of CR or PR or stable disease (SD) based on investigator assessment | up to 26 months
  where best overall response is defined according to RECIST v 1.1, from first treatment administration until the earliest of disease progression, death, or last evaluable tumour assessment before start of subsequent anti-cancer therapy, loss to follow-up or withdrawal of consent
Part 1: Overall survival (OS), defined as the time from treatment start until death from any cause | up to 26 months
Part 1: Change from baseline in EORTC QLQ-C30 physical functioning domain score | at baseline, at month 26
  European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30) The QLQ-C30 is comprised of 30 questions. It incorporates both multi-item scales and single-item measures. These include
  * one global health status/Quality of Life (QoL) scale,
  * five functional scales (physical, role, cognitive, emotional, and social),
  * three symptom scales (fatigue, pain, and nausea and vomiting),
  * and six single items to assess dyspnea, insomnia, appetite loss, constipation, diarrhoea and financial difficulties.
  All scales and single-item measures range in score from 0 to 100.
  * A high score for a functional scale represents a high/healthy level of functioning.
  * A high score for the global health status/QoL represents a high QoL.
  * A high score for a symptom scale/item represents a high level of symptomatology/problems.
Part 1: Change from baseline in EORTC QLQ-C30 role functioning domain score | at baseline, at month 26
Part 1: Occurrence of treatment-emergent AEs leading to study drug discontinuation during the on-treatment period | up to 26 months
Part 2: Duration of objective response (DOR) based on blinded independent central review | up to 27 months
Part 2: Progression-free survival (PFS) based on blinded independent central review | up to 27 months
Part 2: Disease control (DC) based on blinded independent central review | up to 27 months
Part 2: Overall survival (OS), defined as the time from treatment start until death from any cause | up to 27 months
Part 2: Change from baseline in EORTC QLQ-C30 physical functioning domain score | up to 27 months
Part 2: Change from baseline in EORTC QLQ-C30 role functioning domain score | up to 27 months
Part 2: Occurrence of treatment-emergent AEs leading to study drug discontinuation during the on-treatment period | up to 27 months
Part 2: Occurrence of treatment-emergent adverse events (TEAEs) during the on-treatment period | up to 27 months

CONTACTS AND LOCATIONS:
Locations (59):
- United States (16):
  - Infirmary Cancer Care, Mobile, Alabama
  - Mayo Clinic-Arizona, Phoenix, Arizona
  - Valkyrie Clinical Trials, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Virginia Commonwealth University Health- Adult Outpatient Pavilion, Richmond, Virginia
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Bulgaria (2):
  - MHAT UniHospital, Panagyurishte
  - MHAT Heart and brain, Pleven
- China (6):
  - West China Hospital, Sichuan University, Chengdu
  - Sir Run Run Shaw Hospital, Zhejiang University, School of Medicine, Hangzhou
  - Qilu Hospital, Shangdong University, Jinan
  - 960 Hospital of the Chinese People's Liberation Army, Jinan
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - Shanghai Chest Hospital, Shanghai
- France (3):
  - HOP Intercommunal, Créteil
  - Hôpital Cochin, Paris
  - HOP Civil, Strasbourg
- Germany (6):
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Asklepios Fachkliniken München-Gauting, Gauting
  - LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Japan (7):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Sendai Kousei Hospital, Miyagi, Sendai
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Osaka, Sakai
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- Portugal (2):
  - Hospital CUF Descobertas-Lisboa-69316, Lisbon
  - Hospital CUF Porto, Porto
- South Korea (3):
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia
- Taiwan (3):
  - NCKUH, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (4):
  - Leicester Royal Infirmary, Leicester
  - University College Hospital, London
  - The Christie, Manchester
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency